CLINICAL TRIAL: NCT00955136
Title: Utilization of Diagnostic Ultrasound in the Detection and Therapy of Acute Coronary Syndromes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was withdrawn due to many implementation difficulties.
Sponsor: University of Nebraska (Other)
Collaborators: Microvascular Therapeutics, LLC (Industry); The Ruth and Bruce Rappaport Faculty of Medicine (Unknown); Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC) (Other); InCor Heart Institute (Other); Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0286-09-FB
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction
Keywords: ST elevated myocardial infarction; Acute coronary syndrome; MRX 801; Echocardiography
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High MI impulses, myocardial infarction, echocardiography (Experimental): Using the transthoracic three dimensional imaging probe, low mechanical index (MI) will examine wall motion. Intermittent high MI impulses will be administered over the microvasculature where there are wall motion abnormalities using an imaging plan that best aligns itself with the risk area. One vial of MRX 801 to be infused intravenously during echocardiography with high mechanical index impulses.
  Interventions: Device: Use of intermittent high MI impulses during echocardiogram

INTERVENTIONS:
Device: Use of intermittent high MI impulses during echocardiogram — Using the transthoracic three dimensional imaging probe, low mechanical index (MI) will examine wall motion. Intermittent high MI impulses will be administered over the microvasculature where there are wall motion abnormalities using an imaging plan that best aligns itself with the risk area. One vial of MRX 801 to be infused intravenously during echocardiography with high mechanical index impulses.

SUMMARY:
The study will see if mechanical impulses delivered by an echocardiographic probe during a continuous infusion of MRX 801 are capable of improving blood flow in smaller heart vessels in patients with acute coronary syndromes.

DETAILED DESCRIPTION:
Pre-clinical studies have indicated that, during a continuous infusion of intravenous perfluorocarbon-containing microbubbles, the ultrasonic power delivered from a diagnostic ultrasound transducer is capable of restoring microcirculatory flow and improving epicardial recanalization rates following acute coronary thrombotic occlusions. Since both diagnostic ultrasound and intravenous infusions of microbubbles are a Class I indication to assess regional and global left ventricular function and risk area in patients with ST segment elevation myocardial infarction (STEMI), this pilot study will examine whether diagnostic assessments of left ventricular function and risk area size impacts epicardial recanalization rates and infarct size in STEMI.

The aim of this study is to test whether guided high mechanical index impulses from a diagnostic transducer during a continuous infusion of intravenous microbubbles are capable of improving microvascular recanalization and epicardial recanalization rates in STEMI, as assessed by coronary angiography, and recovery of regional microvascular perfusion and function in the post-infarction period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 30 years.
2. Chest Pain occurring lasting less than six hours from onset, and EKG evidence of an acute ST segment elevation myocardial infarction.
3. Arrival in the Emergency Department with above inclusion criteria between 7 am and 7pm.

Exclusion Criteria:

1. Known or suspected hypersensitivity to ultrasound contrast agent used for the study.
2. Complicated hemodynamic instability (i.e., NYHA Class IV heart failure, unstable angina at rest despite medical therapy).
3. Life expectancy of less than two months or terminally ill.
4. Heart transplant recipient, hypertrophic cardiomyopathy, severe valvular disease, acute myo- or pericarditis.
5. Contraindication to Heart Catheterization
6. Known bleeding diathesis or contraindication to glycoprotein 2b/3a inhibitors or aspirin.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07 (Estimated); Primary Completion 2010-01-25 (Actual); Study Completion 2010-01-25 (Actual)

PRIMARY OUTCOMES:
Improved microvascular recanalization and epicardial recanalization rates in STEMI as assessed by coronary angiography and recovery of regional microvascular perfusion and function in the post-infarction period. | 6 weeks
  Improved microvascular recanalization and epicardial recanalization rates in STEMI as assessed by coronary angiography and recovery of regional microvascular perfusion and function in the post-infarction period.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Porter, MD, Principal Investigator — University of Nebraska